CLINICAL TRIAL: NCT00703950
Title: Effects of the Use of a Bottle and a Cup on Breast Sucking Patterns of Premature Infants: Safety and Efficacy
Brief Title: Sucking Pattern of Preterm Infants Using Cup or Bottle Before Breastfeeding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sample size was re- calculated considering sucking pattern parameters
Sponsor: Instituto Fernandes Figueira (Other Government)
Responsible Party: Principal Investigator, Maria Elisabeth Lopes Moreira, MD, Instituto Fernandes Figueira
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAAE-0288.0.008.000-05
Record Dates: First submitted 2008-04-02; First posted 2008-06-24 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Sucking patterns; preterm infants; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1 (Experimental): Cup feeding This is a method to feed preterm babies when breastfeeding is impossible. Feed is provided using cup
  Interventions: Procedure: cup feeding
- A,2 (Active Comparator): bottle feeding - conventional method Bottle feeding is the conventional method to feed preterm infant before breastfeeding or to substitute breastfeeding. We are using this method in the control group.
  Interventions: Procedure: bottle feeding

INTERVENTIONS:
Procedure: cup feeding — Method to feed: cup. This is a method to feed preterm babies when breastfeeding is impossible. Feed is provided using cup
  Other Names: cup method
  Arms: A,1
Procedure: bottle feeding — bottle feeding This is a method to feed preterm babies when breastfeeding is impossible. Feed is provided using bottle
  Other Names: bottle
  Arms: A,2

SUMMARY:
The aim of this study is evaluates the effect of the use of bottle and cup in breast sucking patterns in preterm infants. It will be a randomized blind study. One group will be randomized to use bottle to feed and another one to use a cup to feed. As secondary endpoints, weight gain, days of life to begin full oral feeding, length of hospital stay and breast feeding rates will be observed.

DETAILED DESCRIPTION:
Breastfeeding is the better method to promote adequate growth and development in preterm infants. However, sometimes preterm infants needs to be supplemented with the own mother milk or formula using another methods.

The cup and the bottle have been used in neonatal units, however there is still no evidence to determine the best feeding method, which must be safe, efficient and not jeopardize breast feeding.

The aim of this study is evaluates the effect of the use of bottle and cup in breast sucking patterns. The intervention will be the use of bottle or cup to feed preterm infants before or to supplement breastfeeding after randomization. Nowadays, bottle feeding is the conventional method and we wish to compare sucking patterns after use of bottle or cup. As secondary endpoints, weight gain, days of life to begin full oral feeding, length of hospital stay and breast feeding rates will be observed. In order to achieve this aim, a blind randomized clinical trial will be done with 96 very low birth weight infants, in which a group is randomly selected to be breast fed and get supplementary food using a cup and another to get supplementary food using a bottle.

The trial's inclusion criteria are: birth weight < 1500 g (very low birth weight infants), gestational age from 26 to 32 full weeks, absence of congenital anomalies in the face, head and neck, without severe asphyxia (Apgar < 5 on the 5th minute), negative tests for AIDS, absence of pulmonary chronic disease, mothers willing to breastfeed. Exclusion criteria are: intraventricular hemorrhage (degree III or IV), necrotizing enterocolitis, infection after the beginning of the trial.

Once all newborns in the trial were clinically stable (normal blood pressure without needs of oxygen) and with a volume intake of at least 100 ml/Kg/day of milk through the orogastric tube, they will receive oral-motor stimulation through a stimulation program previously published (2002). Once the newborn meets the criteria to begin oral feeding, an instrumental assessment of non-nutritive sucking and nutritive sucking will be carried out. Intra-oral pressure is assessed in non-nutritive sucking using a pressure monitoring device in a gloved finger: intra-oral negative pressure will be registered using a pressure transducer inserted through a catheter to the tip of the gloved little finger. This catheter will be connected to a second pressure transducer. Simultaneously, breathing (respiratory flow) will be measured using a pneumotachograph coupled to a nasal Prong. Two minutes of sucking will be collected from the moment the newborn responds to the search reflex and grabs the finger. During nutritive sucking assessment, respiration (respiratory flow) will be measured using a pneumotachograph coupled to a nasal Prong. At the same time intra-oral sucking pressure will be recorded by a pressure transducer connected to a catheter located on the mother's breast. Nutritive sucking will take place in the first 5 minutes of breastfeeding. After the first assessment has been concluded, the newborn will be randomly assigned either to the group that will use a cup or a bottle for supplementary feeding using randomized block design. Assessments will be repeated at discharge from the hospital.

The study is taking place at Fernandes Figueira Institute and was approved by the Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* very low birthweight
* gestational age from 26 to 32 complete weeks
* absence of congenital anomalies in the face, head and neck
* absence of severe asphyxia
* negative serology for AIDS
* mothers willing to breastfeed
* absence of pulmonary disease

Exclusion Criteria:

* severe intraventricular hemorrhage
* necrotizing enterocolitis
* infection after the beginning of the trial

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Temporal parameters of sucking | at discharge

SECONDARY OUTCOMES:
days of life at full oral feeding; breastfeeding rates at discharge days of life at full oral feeding breastfeeding rates at discharge | at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabeth l Moreira, PhD, Principal Investigator — Instituto Fernandes Figueira
Locations (1):
- Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro, Brazil